CLINICAL TRIAL: NCT05063981
Title: Biomarkers Evaluation and Effect of Mepolizumab on Lower and Upper Airways Inflammation in Severe Refractory Eosinophilic Asthma
Brief Title: Treatment With Mepolizumab on Patients With Severe Refractory Eosinophilic Asthma
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: University of Palermo (Other); National Research Council (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pascale 09/2020
Record Dates: First submitted 2021-07-15; First posted 2021-10-01 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Severe Eosinophilic Asthma
Keywords: asthma; chronic respiratory disease; mepolizumab; rehabilitation; inflammation
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma; Inflammation | interventions — mepolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, serum, nasal secretions, exhaled breath condensate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe eosinophilic asthma: Patients with severe refractory eosinophilic asthma
  Interventions: Drug: Mepolizumab

INTERVENTIONS:
Drug: Mepolizumab — The effects of treatment with Mepolizumab were evaluated on clinical and laboratory markers of systemic inflammation during a 12 months follow-up period in multiple biological matrices.

SUMMARY:
Understanding how Interleukin-5 blockade modulates both immune and metabolic pathways may clarify the multidimensional impact of biologic therapy in severe eosinophilic asthma. Therefore, this study aimed to assess the impact of mepolizumab on the nasal, bronchial, and systemic metabolomic profiles of consecutive patients with SEA and to explore the associations between these compartment-specific changes and clinical, inflammatory, and functional outcomes.

DETAILED DESCRIPTION:
We conducted a prospective, observational, multicenter cohort study of SEA adult individuals initiating mepolizumab, with 12-month follow-up. Consecutive patients referred to the Pulmonary Rehabilitation Units of the Istituti Clinici Scientifici Maugeri IRCCS in Telese Terme and Tradate, Italy, from September 2021 to September 2023, were screened for eligibility based on the following inclusion criteria: eligibility for mepolizumab treatment according to clinical practice; age between 18 and 75 years; diagnosis of severe eosinophilic refractory asthma, defined as peripheral blood eosinophil count (BEC) > 300 cells/μL and at least two documented exacerbations within the previous 12 months; and ongoing treatment with high daily doses of inhaled corticosteroids (ICS) combined with long-acting β2-agonists (LABA), plus at least one additional controller medication for a minimum of 12 months.

Exclusion criteria included: current smoking; diagnosis of other chronic pulmonary diseases; coexisting chronic rhinosinusitis with nasal polyps; use of systemic corticosteroids at any dose within the 6 weeks prior to enrollment; use of immunosuppressive therapies; receipt of live attenuated vaccines within 30 days prior to enrollment; current or recent history (within the last 5 years) of malignancy, except in cases of complete remission; diagnosis of eosinophilic granulomatosis with polyangiitis (EGPA); upper or lower respiratory tract infections within 30 days prior to signing informed consent or during the screening/run-in period; any clinically significant abnormalities identified during screening through physical examination, vital signs assessment, hematology, or clinical chemistry, which, in the opinion of the investigator, could pose a risk to patient safety or interfere with study outcomes or compliance. Additional exclusion criteria were: known immunodeficiency (primary or secondary); pregnancy; concurrent treatment with other biologics for asthma or other conditions (except for stable allergen immunotherapy, defined as an unchanged dose and regimen at screening); prior biologic therapy for asthma within 6 months before starting mepolizumab; planned surgical procedures during the study period; and participation in another interventional or post-authorization safety study.

The study lasted 24 months, including a 12-month enrollment period followed by a 12-month follow-up. Timepoints at 6 and 12 months were prespecified to capture early consolidation of treatment response and its one-year persistence, in alignment with routine follow up. Prior to inclusion, all participants underwent a clinical examination to assess eligibility. Clinical history was recorded, including age at asthma onset, smoking status, aspirin intolerance, number of exacerbations in the previous year, and asthma control level. Smoking status was recorded as never, former, or current, and current smokers were excluded. Occupational and specific environmental exposures were not systematically collected in this study. Evaluations were performed at baseline (T0), 6 (T6), and 12 months (T12) after initiation of treatment. At each timepoint, respiratory function was assessed and multiple biological matrices were collected to test markers of T2 inflammation and enable metabolomic profiling.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for mepolizumab treatment according to clinical practice;
* age between 18 and 75 years;
* diagnosis of severe eosinophilic refractory asthma, defined as peripheral blood eosinophil count (BEC) > 300 cells/μL and at least two documented exacerbations within the previous 12 months;
* ongoing treatment with high daily doses of inhaled corticosteroids (ICS) combined with long-acting β2-agonists (LABA), plus at least one additional controller medication for a minimum of 12 months.

Exclusion criteria:

* current smoking;
* diagnosis of other chronic pulmonary diseases;
* coexisting chronic rhinosinusitis with nasal polyps;
* use of systemic corticosteroids at any dose within the 6 weeks prior to enrollment;
* use of immunosuppressive therapies;
* receipt of live attenuated vaccines within 30 days prior to enrollment;
* current or recent history (within the last 5 years) of malignancy, except in cases of complete remission;
* diagnosis of eosinophilic granulomatosis with polyangiitis (EGPA);
* upper or lower respiratory tract infections within 30 days prior to signing informed consent or during the screening/run-in period;
* any clinically significant abnormalities identified during screening through physical examination, vital signs assessment, hematology, or clinical chemistry, which, in the opinion of the investigator, could pose a risk to patient safety or interfere with study outcomes or compliance.
* known immunodeficiency (primary or secondary);
* pregnancy;
* concurrent treatment with other biologics for asthma or other conditions (except for stable allergen immunotherapy, defined as an unchanged dose and regimen at screening); prior biologic therapy for asthma within 6 months before starting mepolizumab; planned surgical procedures during the study period;
* participation in another interventional or post-authorization safety study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll patients with severe refractory eosinophilic asthma for whom treatment with mepolizumab is indicated, according to the AIFA recommendations.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Number of exacerbations | Baseline T0; 6 months (T6); 12 months (T12)
  episodes of acute worsening of symptoms
Asthma Control Test (ACT) | Baseline T0; 6 months (T6); 12 months (T12)
  patient self-reported questionnaire, score

SECONDARY OUTCOMES:
Inflammatory markers (Interleukins, TGF-beta, GM-CSF) | Baseline T0; 6 months (T6); 12 months (T12)
  by ELISA test of serum, nasal secretions and exhaled breath condensate, measured as pg/mLof serum
1H-NMR-based metabolomic profiling | Baseline T0; 6 months (T6); 12 months (T12)
  achieved by 1H-NMR spectroscopy of serum, nasal secretions and exhaled breath condensate
peripheral blood eosinophil count (BEC) | Baseline T0; 6 months (T6); 12 months (T12)
  measured by count of cells/uL of blood
Forced expiratory volume (FEV1) | Baseline T0; 6 months (T6); 12 months (T12)
  measured by spirometry, as L
Fractional Exhaled nitric oxide (FeNO) | Baseline T0; 6 months (T6); 12 months (T12)
  measured by an automated electrochemical analyzer (HypAir FeNO), as ppb

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituti Clinici Scientifici Maugeri IRCCS, Telese Terme, BN
  - Istituti Clinici Scientifici Maugeri IRCCS, Tradate, Varese

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Maniscalco M, Ambrosino P, Candia C, Di Stefano A, Gnemmi I, Zappa M, Ambrosino N, Visca D, Motta A. Cytokine and Metabolomic Signatures of Mepolizumab Response Across Upper and Lower Airway Compartments in Severe Eosinophilic Asthma: An Exploratory Analysis. Pharmaceuticals (Basel). 2025 Nov 10;18(11):1704. doi: 10.3390/ph18111704. PMID 41304949
- See also: Pubblication — https://pubmed.ncbi.nlm.nih.gov/41304949/

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-09-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT05063981/Prot_ICF_001.pdf